CLINICAL TRIAL: NCT04446832
Title: VACcination of LIver Transplantation Candidates: Efficacy, Tolerance and Acceptability Prospective Cohort Study.
Brief Title: VACcination of LIver Transplantation Candidates
Acronym: VacLit
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0752
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Liver Transplant; Complications; Vaccination; Complications; Cirrhosis; Chronic Hepatitis
MeSH Terms: conditions — Fibrosis; Hepatitis, Chronic | interventions — Immunogenicity, Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplantation candidates
  Interventions: Other: Vaccine immunogenicity

INTERVENTIONS:
Other: Vaccine immunogenicity — Evaluation of the vaccine immunogenicity by standard approved serological tests

SUMMARY:
Chronic hepatic disease, and especially cirrhosis, are associated to a global dysfunction of the immune system. Liver transplantation represents the only replacement therapy for end-stage liver disease and a curative means of localized hepatocellular carcinoma (HCC) but required immunosuppressive treatment to limit the risk of rejection. Candidates for liver transplantation are at an increased risk for severe infections, some of which can be prevented by vaccination. With regard to vaccine preventable diseases, these patients share the same pitfalls than all immunocompromised individuals: i) a theoretical or proven increased incidence and severity of certain infections warranting specific vaccine recommendations; ii) a decrease in immunogenicity of vaccine; iii) a risk of developing vaccine disease after administration of live attenuated vaccines. It is therefore recommended for all patients awaiting liver transplantation: i) updating the vaccinations recommended in general population (DTPw, MMR); ii) vaccination against viral hepatitis A and B to limit the risk of severe hepatitis; iii) vaccination against pneumococcal infection, influenza and chickenpox more common and more serious in this population. However, these recommendations are based on theoretical assessments and experts opinions; i) immunogenicity of vaccination in cirrhotic patients and persistence of post-transplant protection had been poorly assessed as well as their determinants; ii) there are only a few data regarding the tolerance of vaccinations in this population; iii) vaccination coverage of patients with end-stage liver disease is poorly known in France and; iv) the perception and acceptability of vaccinations have not been evaluated in this population.

Investigators hypothesis is that: the vaccination schedule currently recommended for liver transplantation does not provide adequate protection against vaccine targets 6 months after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* patients waiting for liver transplantation referred by hepato-gastroenterology department as part of the pre-transplant evaluation to the infectiology consultation
* patient who were informed of the study and did not object to participate

Exclusion Criteria:

* patient candidate for multi-organ transplant
* patient who received immunosuppressive therapy, biotherapy and/ or corticosteroid therapy at a dose greater than 10 mg / day of prednisone equivalent for more than 2 weeks within 3 months before vaccination (6 months of rituximab)
* patient who received polyvalent immunoglobulins within the 6 months before the serological evaluation
* patient who received systemic anti-cancer chemotherapy for solid tumor or hemopathy within 6 months preceding the start of vaccination
* splenectomized patients
* asplenic patients for a reason other than liver disease
* chronic infection with the human immunodeficiency virus (HIV)
* patient with any other hereditary immune deficiency or acquired which could compromise the vaccine response or interpretation of serological results
* patient under legal protection measure or unable to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplantation candidates
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of vaccine " responder " according to serological results measured 6 months after liver transplantation | 6 months after liver transplantation
  Vaccine immunogenicity will be assess by titration of specific antibodies by standard approved serological tests and patients will be considered if their antibody title exceed protection threshold defined by the WHO and support by the literature when available (for example for tetanus or diphtheria vaccines), or a 4-fold increase in antibody titers compared to antibodies titers measures before vaccination when a protection threshold is not formally defined (for example for pneumococcus vaccination)

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No